CLINICAL TRIAL: NCT02437032
Title: Type of Gonadotropin During Controlled Ovarian Stimulation Affects the Endocrine Profile in Follicular Fluid and Apoptotic Rate in Granulose Cells
Brief Title: Gonadotropin Type in Ovarian Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Antonio Requena, PhD, MD, IVI Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAD-GV-04-2009-01
Record Dates: First submitted 2014-11-21; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
Keywords: GDF-9; BMP-15; Steroids; Apoptosis rate; Endocrinology
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Urofollitropin; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: recombinant FSH (Active Comparator): An oral contraceptive pill (Microgynon30®, Bayer Hispania, Spain) was taken for a maximum of 21 days, starting on day 1-2 of the menses of the previous cycle. After a wash-period of five days after the last pill, donors started to receive daily doses of 150-300 UI of rFSH (Gonal-F®, Merck-Serono, Spain; n=30) depending on their age, body mass index (BMI) and ovarian response in previous cycles. Daily doses of 0.25 mg gonadotropin- releasing hormone antagonist cetrorelix (Cetrotide®, Merck-Serono, Spain) were started on day six of stimulation in each group. When at least three or more leading follicles reached a mean diameter of ≥18 mm, hCG (Ovitrelle®, 250 µg; Merck-Serono, Spain) was administered subcutaneously
  Interventions: Drug: recombinant FSH
- Group 2:urinary FSH (Active Comparator): An oral contraceptive pill (Microgynon30®, Bayer Hispania, Spain) was taken for a maximum of 21 days, starting on day 1-2 of the menses of the previous cycle. After a wash-period of five days after the last pill, donors started to receive daily doses of 150-300 UI of urinary FSH (uFSH) (Fostipur®, Angelini, Spain; n=30) depending on their age, body mass index (BMI) and ovarian response in previous cycles. Daily doses of 0.25 mg gonadotropin- releasing hormone antagonist cetrorelix (Cetrotide®, Merck-Serono, Spain) were started on day six of stimulation in each group. When at least three or more leading follicles reached a mean diameter of ≥18 mm, hCG (Ovitrelle®, 250 µg; Merck-Serono, Spain) was administered subcutaneously.
  Interventions: Drug: Urinary FSH
- Group 3: with hMG (Active Comparator): An oral contraceptive pill (Microgynon30®, Bayer Hispania, Spain) was taken for a maximum of 21 days, starting on day 1-2 of the menses of the previous cycle. After a wash-period of five days after the last pill, donors started to receive daily doses of 150-300 UI of hMG (HMG-Lepori®, Angelini, Spain; n=30) depending on their age, body mass index (BMI) and ovarian response in previous cycles. Daily doses of 0.25 mg gonadotropin- releasing hormone antagonist cetrorelix (Cetrotide®, Merck-Serono, Spain) were started on day six of stimulation in each group. When at least three or more leading follicles reached a mean diameter of ≥18 mm, hCG (Ovitrelle®, 250 µg; Merck-Serono, Spain) was administered subcutaneously, and transvaginal oocyte retrieval was performed 36 h later.
  Interventions: Drug: hMG

INTERVENTIONS:
Drug: recombinant FSH — Controlled ovarian stimulation with 150-300 UI recombinant FSH
  Other Names: Gonal-F
  Arms: Group 1: recombinant FSH
Drug: Urinary FSH — Controlled ovarian stimulation with 150-300 UI urinary FSH
  Other Names: Fostipur
  Arms: Group 2:urinary FSH
Drug: hMG — Controlled ovarian stimulation with 150-300 UI hMG
  Other Names: hMG-Lepori
  Arms: Group 3: with hMG

SUMMARY:
A key challenge facing reproductive biologists is the integration of the knowledge about oocyte-secreted factors into coherent physiological mechanisms of how oocytes govern folliculogenesis, cumulus cell function, and oocyte and embryo development. Although key oocyte-secreted factors have been identified, understanding their modes of action is complicated by multiple interactions between maternal and oocyte signaling molecules, as well as the constantly changing state of physical interactions between the oocyte and its companion somatic cells during folliculogenesis. Thus, the investigators study aimed to determine if there is any relationship between different gonadotropin preparations and oocyte-secreted factor secretion, the endocrine pattern in follicular fluid, and the apoptotic rate in cumulus cells during controlled ovarian stimulation.

DETAILED DESCRIPTION:
The follicular environment is primarily influenced by the type of gonadotropin the follicle is exposed to during the follicular phase. The role of gonadotropins has been especially important in improving the efficiency of in vitro fertilization. Several studies comparing the use of human menopausal gonadotropin (hMG) with recombinant follicle-stimulating hormone (rFSH) have found significant differences in the endocrinological profile and the follicular dynamics. These differences have been related to the human chorionic gonadotropin (hCG)-driven luteinizing hormone (LH) activity added to hMG. Moreover, differences in the proportion of acid residues in FSH molecules should be considered.

On the other hand, the main physiological regulatory hormones of follicular survival are the gonadotropins. Suppression of serum gonadotropins leads to massive apoptosis of granulosa cells in developing follicles resulting in atresia; whereas, gonadotropin treatment of early antral and pre-ovulatory follicles prevents this unplanned apoptosis. However, studies using cultured rat granulosa cells have shown that treatments with FSH or LH/hCG are ineffective in preventing spontaneous apoptosis, suggesting neighboring theca cells and local factors produced in the ovary are important for regulation of follicle growth and atresia.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* regular menstrual cycles
* no hereditary or chromosomal diseases normal karyotype negative for sexually transmitted diseases
* at least seven antral follicles per ovary

Exclusion Criteria:

* PCO

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
GDF-9 and BMP-15 secretion | 3 years
  To measure GDF-9 (ng/ml) and BMP-15 (micrograms/microliter)

SECONDARY OUTCOMES:
Steroids levels in follicular fluid (estradiol, progesterone, testosterone, FSH) | 3 years
  To measure estradiol (pg/ml), progesterone (ng/ml), FSH (mUI/ml) and testosterone (ng/ml)
Apoptotic rate in cumulus cells | 3 years
  To measure early and late apoptotic rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Requena, PhD, MD, Principal Investigator — IVI Madrid

REFERENCES:
- [Result] Gilchrist RB, Lane M, Thompson JG. Oocyte-secreted factors: regulators of cumulus cell function and oocyte quality. Hum Reprod Update. 2008 Mar-Apr;14(2):159-77. doi: 10.1093/humupd/dmm040. Epub 2008 Jan 5. PMID 18175787
- [Result] Smitz J, Andersen AN, Devroey P, Arce JC; MERIT Group. Endocrine profile in serum and follicular fluid differs after ovarian stimulation with HP-hMG or recombinant FSH in IVF patients. Hum Reprod. 2007 Mar;22(3):676-87. doi: 10.1093/humrep/del445. Epub 2006 Nov 16. PMID 17110397
- [Result] Orisaka M, Orisaka S, Jiang JY, Craig J, Wang Y, Kotsuji F, Tsang BK. Growth differentiation factor 9 is antiapoptotic during follicular development from preantral to early antral stage. Mol Endocrinol. 2006 Oct;20(10):2456-68. doi: 10.1210/me.2005-0357. Epub 2006 Jun 1. PMID 16740654